CLINICAL TRIAL: NCT06166537
Title: Graduated Compression Stocking as an Adjunct to Extended Duration Pharmacological Thromboprophylaxis for Venous Thromboembolism Prevention
Brief Title: GRACE: Evaluating Compression Stockings in Patients That Require Extended Duration Pharmacological Thromboprophylaxis
Acronym: GRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22HH7932
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Venous Thromboembolism; Surgery
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: Assessor-blinded randomised controlled trial with a non-inferiority comparison
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDPTP plus GCS (Other): Control - Extended duration pharmacological thromboprophylaxis (EDPTP) and Graduated compression stockings (GCS).
  Interventions: Other: Graduated compression stockings
- EDPTP alone (Other): Intervention - Extended duration pharmacological thromboprophylaxis (EDPTP) alone, no stockings
  Interventions: Other: No Graduated compression stockings

INTERVENTIONS:
Other: Graduated compression stockings — Graduated compression stockings are standard care (control)
  Other Names: TED Stockings
  Arms: EDPTP plus GCS
Other: No Graduated compression stockings — No Graduated compression stockings is the intervention
  Other Names: No TED Stockings
  Arms: EDPTP alone

SUMMARY:
Individuals attending the hospital to undergo operations are at risk of developing blood clots in the legs, known as deep vein thrombosis (DVT). A clot in the leg can cause swelling, pain, and other long-term problems. If a clot in the leg breaks off and travels to the lungs, it can cause problems with the lungs' ability to move oxygen from the air into the blood and may be life-threatening. This is known as pulmonary embolism (PE). DVT and PE are known collectively as venous thromboembolism or VTE.

The importance of preventing VTE in surgical patients is widely recognised, with two main strategies used: thinning the blood with regular injections and/or tablets and wearing elastic stockings to help stop blood from sitting in the leg veins where it can clot.

Evidence for using elastic stockings to prevent VTE has recently been challenged. Additionally, there is a lack of evidence for the additional benefit of stockings over and above that of blood thinning medications. If stockings were to reduce VTE over and above blood thinning medication, these benefits need to be weighed against the risks and disadvantages of stockings, including discomfort, restricting blood flow to the leg causing blisters and wounds in addition to the cost. If stockings were found not to reduce the risk of clots, they would no longer need to be used in these patients, thus reducing the disadvantages of stockings, and saving the NHS millions of pounds per year.

Certain types of operations (300,000 per year in the UK) are linked with a particularly high risk of VTE, including cancer surgery, surgery in the abdomen and pelvis, and bone (orthopaedic) surgery. In these cases, patients are offered blood thinning medications both during their hospital stay and for a period after they have left the hospital. Furthermore, these patients are offered stockings to wear while in the hospital.

It is not known if, in patients who receive blood thinning medications both in hospital and after discharge, the addition of wearing stockings whilst in hospital reduces their risk of VTE any further.

The purpose of this study is to investigate if it is worthwhile using stockings, in addition to blood thinning medication, to reduce blood clots after surgery. People enrolled in the study will be those at the highest risk of VTE and require an extended period of medication to reduce the risk of a blood clot.

A computer will randomly choose one of the below treatments by chance to make the trial fair:

A) Extended duration clot-reducing medicine in addition to stockings B) Extended duration clot-reducing medicine alone

The surgery and all the other medical care will continue as normal. Everyone in the study will get an ultrasound scan at 21 - 35 days after their operation to check if they have developed a blood clot. This is an additional scan, not routinely performed in the NHS, to make sure that all blood clots are detected at an early stage. Participants will receive a phone call at 7, 21-35 and 90 days after their treatment to see if they have developed a blood clot or had any problems with the treatment.

DETAILED DESCRIPTION:
Research question: Is it beneficial to provide graduated compression stockings (GCS) in addition to extended duration pharmacological thromboprophylaxis (EDPTP) for surgical patients at highest risk of venous thromboembolism (VTE)? Background: Hospital-acquired thrombosis (HAT) is defined as any VTE within 90 days of hospital admission, encompassing both deep vein thrombosis (DVT) and pulmonary embolism (PE). HAT represents a significant cause of preventable mortality, with over 12,000 people dying each year from hospital-associated VTE in the UK, 10-fold higher than the number dying from road traffic accidents.

Previous studies report that the risk of untreated high-risk surgical patients developing HAT is as high as 40-60% in orthopaedic patients and 15-40% in general surgery patients. For these patients at highest risk of VTE, key prevention strategies include extended pharmacological thromboprophylaxis (EDPTP) prescribed beyond hospital discharge and provision of graduated compression stockings (GCS). There is compelling evidence to support the use of pharmacological thromboprophylaxis, however, there is little evidence to support the use of additional GCS alongside causing complications in as many as 5% of patients. The cost of providing GCS equates to a minimum of £31.05 per patient episode, with as many as 270,000 relevant procedures conferring a high-risk of VTE, it could be costing the NHS £8.3 million per annum.

Aims and objectives: The GRACE trial aims to establish whether:-

1. patients undergoing surgical procedures requiring EDPTP benefit from additional GCS to prevent VTE
2. patients receiving GCS experience an increased rate of adverse events

Methods: Assessor-blinded randomised controlled trial with a non-inferiority comparison. 8,608 participants will be randomised in a 1:1 fashion to one of two thromboprophylaxis strategies:

1. EDPTP* in addition to GCS, or
2. EDPTP alone *EDPTP includes any anti-thrombotic agent prescribed at a prophylactic dose for prevention of VTE, including low-molecular weight heparin, directly acting oral anticoagulants, or antiplatelet therapy.

Everyone in the study will get an ultrasound scan at 21 - 35 days after their operation to check if they have developed a blood clot. This is an additional scan, not routinely performed in the NHS, to make sure that all blood clots are detected at an early stage. Participants will receive a phone call at 7, 21-35 and 90 days after their treatment to see if they have developed a blood clot or had any problems with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age)
* Participants undergoing elective surgery; risk assessed as requiring EDPTP

Exclusion Criteria:

* Contraindications to EDPTP or GCS
* Individuals requiring therapeutic anticoagulation e.g., anticoagulation for previous DVT
* Known thrombophilia or thrombogenic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8608 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Imaging-confirmed lower limb Deep Venous Thrombosis with or without symptoms, or Pulmonary Embolism with symptoms. | up to 90 days post-surgery
  The number of participants that have a Venous thromboembolism (VTE) event.

SECONDARY OUTCOMES:
Mortality | up to 90 days post-surgery
  The number of participants that die
Adverse event | up to 90 days post-surgery
  The number of participants that experience adverse events related to GSC or EDPTP
Safety outcomes | up to 90 days post-surgery
  The number of participants that experience major bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - North Bristol NHS Trust, Bristol
  - Imperial College Healthcare NHS Trust, London
  - University College London NHS Trust, London

IPD SHARING:
Plan to Share IPD: No